CLINICAL TRIAL: NCT02562729
Title: A Simplified Approach of Complete Nerve-sparing Type C1 Radical Hysterectomy for Cervical Cancer, a Phase II Study
Brief Title: Complete Nerve-Sparing Radical Hysterectomy for Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zsfdu-obgyn-003
Record Dates: First submitted 2015-09-18; First posted 2015-09-29 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-07

CONDITIONS: Cervical Squamous Cell Carcinoma; Cervical Adenocarcinoma; Malignant Neoplasm of Cervix Stage IB1; Stage IIA1 Cervical Cancer
Keywords: Cervical cancer; Nerve-sparing hysterectomy; simplified
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nerve-Sparing Radical Hysterectomy (NSRH) (Experimental): Type C1 Hysterectomy
  Interventions: Procedure: Nerve-Sparing Radical Hysterectomy

INTERVENTIONS:
Procedure: Nerve-Sparing Radical Hysterectomy — Type C1 NSRH Removal indwelling catheter on day 4 after surgery
  Other Names: Fully Pelvic-Nerve Plexus Preserved

SUMMARY:
The purpose of this study is to evaluate the feasibility of complete nerve-sparing type C1 radical hysterectomy in cervical cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the rate of postvoid residual urine volume (PVR) <50ml on postoperative day 4 in patients with stage IB1 and IIA1 cervix cancer underwent complete nerve-sparing type C1 radical hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years to <= 70 years.
* Women with histologically confirmed, primary adenocarcinoma or squamous cell carcinoma of the uterine cervix.
* Stage IIA1, or IB1 disease.
* Karnofsky performance status >70.
* Patients who comply with follow-up.
* With written informed consent.

Exclusion Criteria:

* Age>70
* History of lower urinary tract damage or surgery.
* With abnormal urodynamic study results.
* Karnofsky performance status <70.
* Patients who have uncontrolled psychological disorders.
* Unwilling to or unable to comply with protocol.
* Prior treatment with pelvic radiotherapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with fully pelvic nerve plexus preserved | up to 30 days
  Proportion of patients who had a postvoid residual urine volume (PVR) under 50ml at postoperative day 4
Proportion of patients removing indwelling catheter | up to 30 days

SECONDARY OUTCOMES:
The rate of 36-month local control | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Rongyu Zang, MD,PhD, Principal Investigator — Fudan University Shanghai Zhongshan Hospital
Locations (1):
- Fudan University Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang Y, Shi T, Yin S, Ma S, Shi D, Guan J, Xiang L, Liu Y, Ren Y, Tan D, Zang R. An improved nerve-sparing radical hysterectomy technique for cervical cancer using the paravesico-vaginal space as a new surgical landmark. Oncotarget. 2017 Jul 5;8(52):90413-90420. doi: 10.18632/oncotarget.19011. eCollection 2017 Oct 27. PMID 29163840